CLINICAL TRIAL: NCT06612684
Title: A New Syndesmotomy Technique for Tooth Extractions: Preserving the Integrity of the Alveolar Bone
Brief Title: A New Syndesmotomy Technique for Tooth Extractions to Preserve the Alveolar Bone
Acronym: SINDESM-EXt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Manicone Paolo Francesco, Associate professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6139
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Tooth Extraction; Piezoelectric Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Piezoelectric syndesmotomy of single-rooted teeth (Experimental): Patients who need the extraction of a single-rooted hopeless tooth will be included in the intervention arm. The extraction of the tooth will be executed by piezoelectric syndesmotomy and by the use of forceps.
  Interventions: Device: Piezoelectric syndesmotomy

INTERVENTIONS:
Device: Piezoelectric syndesmotomy — Syndesmotomy, the first phase of tooth extraction, will be provided by a piezoelectric device instead of manual instruments.

SUMMARY:
In both surgical and nor surgical tooth extractions, the first phase is done by syndesmotomy. This procedure allows to interrupt the fibers of the periodontal ligament. Traditionally, syndesmotomy is done by manual instruments. Usually, the manual approach leads to the loss of the vestibular cortical plate due to the size of those instruments.

The piezoelectric surgery device provides an alternative to manual instruments. Its advantages are: selectivity for hard tissues; better cut control; protection of soft tissue, vessels and nerves; post-op pain and discomfort reduction.

The aim of this study is to evaluate a piezosurgery driven syndesmotomy technique during tooth extraction.

DETAILED DESCRIPTION:
Piezoelectric bone surgery is a recent and innovative technology, permitting a selective cut of mineralized tissue while sparing soft tissue. Similar to a dental scaler, a high frequency vibration, in the range of 25-35 kHz, is transmitted to a metallic tip. The handpiece of the instrument is equipped with a sterile irrigation system and light-emitting diode (LED) light, which improves visibility and overall safety. Piezoelectric surgery is particularly useful when performing delicate bone procedures such as periodontal or endodontic surgery. It is also indicated when performing more invasive bone surgery such as maxillectomy, mandibulectomy, and condylectomy, where preservation of neurovascular structures is important. Piezoelectric surgery is still employed in tooth extraction of third lower molars. In literature, there are low evidence of the use of piezoelectric surgery for single-rooted tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Single-rooted tooth to extract that:
* has mobility grade 0 or 1
* is considered hopeless or needs to be extracted due to orthodontic indication
* Sign of informed consent

Exclusion Criteria:

* Age lower than 18 years old
* Pregnancy
* Heavy smokers (more than 10 cigarettes a day)
* Uncompensated systemic diseases
* Drugs that influence wound healing (radiotherapy in the last year, bisphosphonates)
* Low compliance due to psychiatric diseases
* Mobility grade 2 or 3
* Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean difference of bone sounding (mm) before and after tooth extraction | Day0, before and after the surgical extraction
  Bone sounding is a measurement in millimeters that represents the distance between alveolar crest and free gingival margin. This measurement is taken under local anesthesia before and after the tooth extraction.
  This outcome provides informations about the integrity of the alveolar bone before and after the surgical procedure.
  Six sites for tooth are considered. The mean difference expressed in millimeters is considered for each site.

SECONDARY OUTCOMES:
Post-operative pain evaluation: VAS scale value (0-10) at D1, D3, D7 and D21 | Day 1, 3, 7, 21 after tooth extraction
  The Visual Analog Scale (VAS SCALE - score 0-10) is submitted to the patient after tooth extraction to evaluate the post-operative pain and discomfort in four different times after the surgical procedure.
Post-operative pain trend evaluation: VAS scale values difference (0-10) at D1, D3, D7 and D21 | Day 1, 3, 7, 21 after tooth extraction
  The Visual Analog Scale (VAS SCALE - score 0-10) is submitted to the patient after tooth extraction to evaluate the post-operative pain and discomfort in four different times after the surgical procedure. The trend of VAS value at each time is observed
Post-operative quality of life evaluation: QoL score (0-100) at D1, D3, D7 and D21 | Day 1, 3, 7, 21 after tooth extraction
  The Quality of Life score (QoL score - score 0-100) is submitted to the patient after tooth extraction to evaluate the post-operative quality of life in four different times after the surgical procedure.
Post-operative quality of life trend evaluation: QoL score differences (0-100) at D1, D3, D7 and D21 | Day 1, 3, 7, 21 after tooth extraction
  The Quality of Life score (QoL score - score 0-100) is submitted to the patient after tooth extraction to evaluate the post-operative quality of life in four different times after the surgical procedure. The trend of QoL value at each time is observed
Number of analgesics taken a week after the surgical procedure | From surgical procedure to day 7
  It is asked to each patient how many analgesics he needed after the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: PAOLO FRANCESCO MANICONE, Associate professor, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No